CLINICAL TRIAL: NCT03264508
Title: Passive Heat Therapy and Age-associated Physiological Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Seals (Other)
Responsible Party: Sponsor-Investigator, Douglas Seals, Professor of Distinction, University of Colorado, Boulder
Organization: University of Colorado, Boulder (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-0757
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Aging
Keywords: endothelial function; arterial stiffness; heat; hot water immersion
MeSH Terms: interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: Randomized, controlled (parallel design), single-blind
Who Masked: Investigator
Masking Description: Investigators collecting and analyzing data will be blinded to subject treatment arms. It is not possible to blind subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat therapy (Experimental): Hot water immersion 3-4x per week for 8-10 weeks
  Interventions: Behavioral: Heat therapy
- Thermoneutral water immersion (Sham Comparator): Thermoneutral water immersion 3-4x per week for 8-10 weeks
  Interventions: Behavioral: Thermoneutral water immersion

INTERVENTIONS:
Behavioral: Heat therapy — 30 sessions (3-4x per week for 8-10 weeks) of hot water immersion in 40°C water, sufficient to raise body core temperature to 38.5°C.
  Arms: Heat therapy
Behavioral: Thermoneutral water immersion — 30 sessions (3-4x per week for 8-10 weeks) of hot water immersion in 36°C water to prevent changes in body core temperature >0.2°C.
  Arms: Thermoneutral water immersion

SUMMARY:
This study aims to determine the effects of 8-10 weeks of repeated hot water immersion ("heat therapy") vs. thermoneutral water immersion on vascular function in late middle-aged to older (55-79 years) adults.

DETAILED DESCRIPTION:
Advancing age is the primary risk factor for cardiovascular diseases (CVD), which remain the leading cause of death in the developed world. The key process that links aging to increased risk of CVD is the development of arterial dysfunction, including impaired endothelial function and arterial stiffening. In addition, age-associated impairments in arterial function have been linked to other diseases/disorders of aging, including cognitive impairments, Alzheimer's disease and dementia, and motor disorders/disability.

Passive heat therapy, in the form of repeated use of hot baths and saunas, has been used by several cultures for centuries; however, the physiological benefits are only now being elucidated. For example, recent studies have found that lifelong habitual sauna use is associated with considerably reduced risk of all-cause mortality, sudden cardiac death, CVD-related death, and Alzheimer's disease and dementia. In addition, 8-10 weeks of hot water immersion in young adults has been shown to improve endothelial function and reduces arterial stiffness and blood pressure. Therefore, the investigators expect heat therapy to similarly improve vascular function, as well as cognitive and motor function, in middle-aged to older adults who are at greater risk of CVD and related diseases/disorders.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent.
* Aged 55-79 years. Women must be postmenopausal and not taking hormone replacement therapy within the past year.
* Sedentary to recreationally active: participating in vigorous aerobic exercise <4x/wk for ≥ 3 yrs.
* Able to refrain from the use of dietary supplements, anti-inflammatory medications, and prescription medications for 24-48h prior to experimental testing.
* Generally healthy (no overt clinical disease), as determined by medical history, physical examination, blood and urine chemistries.
* Ankle-brachial blood pressure index >0.7
* Total cholesterol <240 mg/dl (<6.2 mmol/L)
* Fasting plasma glucose <126 mg/dl (<7.0 mmol/L)
* Systolic blood pressure < 160 mmHg and >100 mmHg
* Glomerular filtration rate > 60 ml/min/1.73 m2
* Mini mental state exam score > 20 points
* Body mass index (BMI) <30 kg/m2
* Weight stable in the prior 3 months (≤ 2 kg weight change) and willing to remain weight stable over the course of the study
* Free from alcohol dependence or abuse, as defined by the American Psychiatry Association, Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).

Exclusion Criteria:

* Current use of certain prescription medications that may interfere with thermoregulation and/or blood pressure control during heat stress. These include anti-hypertensives (in particular beta-blockers), nitrates and nitrites (e.g. nitroglycerin), PDE5 inhibitors (e.g. Viagra), anticholinergics (e.g. amitriptyline), and alpha-blockers (e.g. Flomax).
* Orthostatic hypotension
* Current or past smoking within the last 5 years
* Recent major change in health status within previous 6 months (i.e. surgery, significant infection or illness).
* Chronic clinical diseases (e.g., inflammatory bowel diseases/irritable bowel syndrome, coronary artery/peripheral artery/cerebrovascular diseases, diabetes, chronic kidney disease requiring dialysis, neurological disorders or diseases that may affect motor/cognitive functions [multiple sclerosis, Parkinson's disease, polio, Alzheimer's disease, dementia or other brain diseases of aging]).
* History of heat-related illness
* Open wounds or skin lesions. History of skin-related conditions or sensitivities to prolonged water immersion or exposure to pool chemicals.
* Blood donation within the past 2 months
* Inability to tolerate blood draws, intravenous catheters, and/or fingertip blood sampling, including past fainting in response to blood sampling.
* Rectal, anal, vaginal, or prostate surgery within the last 6 months, current or recent (within the last 6 months) hemorrhoids, or related concerns regarding use of rectal thermistor

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | 0 and 8 weeks
  Measure of endothelial function
Carotid-femoral pulse wave velocity | 0 and 8 weeks
  Measure of central arterial stiffness
Mean arterial blood pressure | 0 and 8 weeks
  Brachial artery blood pressure, measured in triplicate (and averaged) following 20 min of supine rest

SECONDARY OUTCOMES:
Cerebrovascular reactivity | 0 and 8 weeks
  Measure of cerebral vascular function; magnitude of increase in blood flow through the middle cerebral artery in response to breathing 5% CO2
Fluid cognition composite score | 0 and 8 weeks
  Multiple domains of cognitive function (incl. executive function, memory, processing speed) assessed using the NIH toolbox (aggregated into one reported value)
Motor function composite score | 0 and 8 weeks
  Multiple domains of motor function (incl. endurance, strength, dexterity) assessed using the NIH toolbox (aggregated into one reported value)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Seals, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunt VE, Howard MJ, Francisco MA, Ely BR, Minson CT. Passive heat therapy improves endothelial function, arterial stiffness and blood pressure in sedentary humans. J Physiol. 2016 Sep 15;594(18):5329-42. doi: 10.1113/JP272453. Epub 2016 Jun 30. PMID 27270841